CLINICAL TRIAL: NCT05888701
Title: "Don't Eat me" Signal in Hematological Malignancies: CD24 as New Target to Improve Anti-cancer Immunity.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: CD24.DEM
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Mantle-cell Lymphoma; B Cell Chronic Lymphocytic Leukemia
Keywords: MCL; NHL; CLL; TAM
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — peripheral blood and bone marrow blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mantle-cell Lymphoma (MCL) is a B-cell non-Hodgkin's lymphoma (NHL) with heterogeneous behavior,ranging from indolent phenotype to highly aggressive and drug resistant cases with dismal prognosis.Disease progression and drug resistance may be generated by Tumor Microenvironment (TME),owing that M2-like immunosuppressive tumor associated macrophages (TAM) are pathologically functional in providing survival signals to MCL cells-and TME is known to help mask tumoral cells from host immune system.Similarly, Chronic Lymphocytic Leukemia (CLL) is a B-cell malignancy characterized by increased circulating number of mature B lymphocytes that eventually reside into bone marrow and lymphoid tissues as well.Higher number of circulating abnormal B cells is secondary to a balance between increased proliferation and decreased apoptosis activities,sustained by signals also deriving from TME.As a matter of fact,TME harbors different cell compounds and monocyte-derived Nurse-like cells (NLCs) resemble the M2-like macrophage immunosuppressive profile and turned out to be an important component able to interact with CLL cells, providing improvement of proliferation and survival.Recently, cancer-expressed CD47 was found to be involved in tumor immune escape through interaction with Signal Regulatory Protein-α (SIRP-α) expressed by TAM,being able to quench phagocytosis. Interestingly,"Don't Eat Me" signal (DEMs) blockade with anti-CD47 monoclonal Antibody (mAb) showed promising activity in pretreated NHL,through increase of phagocytosis by TAM.CD24 was also demonstrated to be involved in DEMs in solid cancer.As a matter of fact, tumor-expressed CD24 promotes immune evasion through its interaction with the inhibitory receptor sialic-acid-binding Ig-like lectin10 (Siglec-10),expressed by TAM with immunosuppressive phenotype (M2-like).In a preclinical model of CD24+ solid tumors (ovarian and breast cancer) the blockade of CD24-Siglec-10 interaction with anti-CD24 mAb showed improvement of TAM-associated phagocytosis in vitro and TAM-dependent reduction of tumor growth and increase of survival in vivo.It is worth mentioning that CD24 can be expressed in some phases of B-cell differentiation and both MCL and CLL derives from a B-cell precursor with upregulated CD24.In this setting,CD24 might play a critical role in the anti-phagocytic signal, since MCL and CLL represents a subset of B-cell malignancies with a considerable hostile TME with M2-like TAM,able to jeopardize anti-cancer immunity.Therefore, the possibility to boost innate anti-cancer immunity through this DEMs blockade could provide new therapeutic options to previous heavily pretreated relapsed/refractory MCL and CLL patients.

DETAILED DESCRIPTION:
MCL is an aggressive B-NHL with dismal prognosis with high probability of relapse after conventional immunochemotherapeutic regimen. CLL is instead an incurable chronic B-cell malignancy with higher probability of relapse after several lines of conventional therapies and a non-negligible risk of progression into an aggressive lymphoma. Further approaches are needed to provide valid alternatives for these relapsed and refractory diseases. In these two settings, TME is known to be involved in cancer cell survival and confers a negative impact on standard treatment efficacy and adoptive T cell immunity, for which new immunotherapeutic agents could be an alternative approach in case of poor prognostic settings. Within TME, TAM are involved in improving tumor growth survival in MCL and CLL, dampening immunotherapy as well. Anti-CD47 mAb turned out to be a consistent DEMs that, once blocked, is able to improve phagocytosis and clearance of tumor cells in blood cancer. CD24 has been recently validated as another DEMs in preclinical analysis in solid cancer. Since CD24 is expressed during early phase of B-cell differentiation, MCL and CLL might take advantage of the blockade of this signal, since TAM and NCLs are strictly interconnected with their corresponding tumoral cells, providing tumor cell proliferation and immune escape.

To fulfill the purposes of this project, collection of leftover patient-derived samples will be routinary performed at the time of diagnosis and at the time of relapse of the disease, in this latter case with the aim to check any CD24, CD47 and CD20 surface expression modification on B-cell blasts (e.g., clone selection with CD24/CD47 upregulation after conventional regimen), SIRP-α and Siglec-10 expression on patient-derived Monocyte/Macrophage system (expressing higher levels of DEMs ligands as potential mechanism of resistance after conventional therapy).

Furthermore, phagocytosis assays with samples obtained at the time of relapse will be compared with the equivalent experiments performed with the samples collected at the time of diagnosis to evaluate any potential differences.

As previously described, phagocytosis analysis will be based on a co-culture process that involves the use of the anti-CD24 antibody (alone or in combination with other antibodies described in the secondary endpoint) incubating with macrophages (from healthy donor or from patient) and patient tumor cells (MCL or CLL), this latter labeled with a fluorescent substance (i.e., CFSE). Macrophage staining (with anti-CD11b-PE antibody) and subsequent flow cytometric analysis will be performed: the ratio between double stained macrophages (CD11b-PE+/CFSE+) and single stained macrophages (CD11b-PE+) will provide the entity of phagocytosis, which will be compared with the negative control and the other experimental conditions (antibody combinations described later in the secondary endpoints). The double staining of macrophages provides indirect results of phagocytosis (if the macrophage phagocytes CFSE+ cells, it will also acquire this staining in addition to that due to the anti-CD11b-PE antibody).

Finally, donor-derived macrophages will be isolated from PBMC obtained from leftover peripheral blood which remained within the circuit used for plateletpheresis of healthy donors. As a matter of fact, residual blood (almost 15 ml) can be found in the reservoir of this circuit that is normally trashed after the procedure. Donors will sign informed consent for use of leftover material for research purposes and this project in particular.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria:

* Signed and dated EC-approved informed consent
* Diagnosis of Mantle-cell Lymphoma (MCL) or B-cell Chronic Lymphocytic Leukemia (CLL) defined according to World Health Organization (WHO) criteria.
* Female or male, 18 years of age or older.
* ECOG performance status 0-3.
* Willingness and ability to comply with routine clinical practice and study procedures.

Donors inclusion criteria:

* Signed and dated EC-approved informed consent.
* Healthy volunteers agreed to undergo plateletpheresis.
* Female or male, 18 years of age or older.
* Willingness and ability to comply with Transfusion Medicine clinical practice and study procedures.

Exclusion Criteria

Patient exclusion criteria:

* Other hematological diseases defined by WHO criteria different from MCL and CLL.
* Previous treatment regimens that included allogeneic stem cell transplantation (ASCT).

Donors exclusion criteria:

-Healthy volunteers agreed to perform any kind of donations with the exception of plateletpheresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This single-center will enroll approximately 30 patients suffering from MCL (n=10) and CLL (n=20) referred to the Department of Hematology at San Gerardo Hospital, Monza, Italy.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Primary endopoint | 36 months
  Rate of phagocytosis of human M2-like macrophages co-cultured with MCL and CLL blast cells treated with anti-CD24 mAb.

SECONDARY OUTCOMES:
Secondary endopoints | 36 months
  * Rate of phagocytosis with patient-derived monocytes system and autologous MCL/CLL blast cells with anti-CD24 mAb.
  * Rate of phagocytosis with different mAb combinations and statistical comparison (anti-CD24, anti-CD47, anti-CD20, anti-CD24+anti-CD47, anti-CD47+anti-CD20, anti-CD24+anti-CD20, anti-CD47+anti-CD24+anti-CD20 mAbs) for donor-derived and patient-derived human macrophages co-cultured with human MCL and CLL blast cells derived from patients.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Aroldi, Principal Investigator — Ospedale San Gerardo - ASST Monza
Locations (1):
- Andrea Aroldi, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: No